CLINICAL TRIAL: NCT01405924
Title: EMEND® IV In Salvage Treatment of Chemotherapy-Induced Vomiting
Brief Title: Fosaprepitant (MK-0517, EMEND® IV) In Salvage Treatment of Chemotherapy-Induced Vomiting (MK-0517-030)
Acronym: EVADE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0517-030
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — fosaprepitant; Aprepitant; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fosaprepitant 150 mg (Experimental): Women with breast cancer receiving anthracycline-cyclophosphamide (AC)-like chemotherapy and women with gynecological cancer receiving carboplatin-paclitaxel (CT) chemotherapy receive fosaprepitant 150 mg administered intravenously (IV) on Day 1 of Cycle 2 of chemotherapy
  Interventions: Drug: Fosaprepitant dimeglumine; Drug: 5-HT3 RA; Drug: Dexamethasone; Drug: Rescue medication

INTERVENTIONS:
Drug: Fosaprepitant dimeglumine — Fosaprepitant 150 mg, IV on Day 1 of chemotherapy in Cycle 2
  Other Names: MK-0517, EMEND® IV
Drug: 5-HT3 RA — 5-HT3 RA will be administered at the same dosage in Cycle 2 of chemotherapy as was used for each particpant in Cycle 1 of chemotherapy.
Drug: Dexamethasone — Dexamethasone will be administered at the same dosage in Cycle 2 of chemotherapy as was used for each particpant in Cycle 1 of chemotherapy.
Drug: Rescue medication — Rescue medication is defined as any medication used to relieve the symptoms of established nausea or vomiting. Multiple medications are permitted by the protocol and may be taken by the participant, including 5-HT3 antagonists, phenothiazines and benzodiazepines.

SUMMARY:
This study will assess the efficacy of a single dose of intravenous (IV) fosaprepitant (MK-0517, EMEND® IV) as salvage therapy when added to a 5-hydroxytryptamine receptor 3 antagonist (5-HT3 RA) and dexamethasone for the prevention of chemotherapy-induced vomiting (CIV) in participants who experienced CIV in the first cycle of moderately emetic chemotherapy (MEC). The primary hypothesis is that there will be no vomiting and no retching in at least 20% of participants during the second cycle of MEC in participants who previously experienced vomiting during the first cycle of MEC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either breast or gynecological cancer
* Receiving either AC-like or CT MEC
* Experienced at least 1 episode of vomiting or retching during the first 5 days following Cycle 1 of chemotherapy that was thought to be due to chemotherapy. Received standard chemotherapy-induced nausea and vomiting (CINV) prophylaxis not containing aprepitant or fosaprepitant
* No change in chemotherapy at Cycle 2
* No change in Cycle 1 antiemetic regimen at Cycle 2
* Eastern Cooperative Oncology Group (ECOG) status 0-1

Exclusion Criteria:

* Requires increase in systemic corticosteroid therapy
* Used benzodiazepines or opiates in the 48 hours prior to Cycle 2 chemotherapy
* Received or will receive radiation therapy to the abdomen or pelvis in the week prior to Visit 1 or in Days 1-6 following chemotherapy
* Vomited in the 24 hours prior to Treatment Day 1
* Pregnant or breast-feeding
* Participating in a study with aprepitant or fosaprepitant or has taken an investigational drug in the last 4 weeks
* Symptomatic central nervous system metastasis
* History of other malignancies in the last 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2013-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0517-030&kw=0517-030&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fosaprepitant 150 mg
Started | 111
Completed | 101
Not Completed | 10
Not completed — Protocol Violation | 8
Not completed — Missing/Incomplete Data | 2

BASELINE CHARACTERISTICS:
Groups:
- Fosaprepitant 150 mg: Women with breast cancer receiving AC-like chemotherapy and women with gynecological cancer receiving CT chemotherapy receive fosaprepitant 150 mg administered IV on Day 1 of Cycle 2 of chemotherapy
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.83 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Vomiting and No Retching During Cycle 2 of Chemotherapy
Description: A vomiting episode is defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes are separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. The percentage of partcipants with no vomiting and no retching episodes 0-120 hours following chemotherapy in Cycle 2 was calculated.
Time Frame: Up to 120 hours following initiation of chemotherapy in Cycle 2
Population: The population consisted of all participants who received chemotherapy, received a dose of study drug, had no protocol deviations and had complete data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 101
Percentage of Participants | 57.43

2. Secondary Outcome: Percentage of Participants With No Vomiting and No Retching During Cycle 2 of Chemotherapy Per Type of Chemotherapy
Description: A vomiting episode is defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes are separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. The percentage of partcipants with no vomiting and no retching episodes 0-120 hours following initiation of chemotherapy in Cycle 2 was calculated based on type of chemotherapy received.
Time Frame: Up to 120 hours following initiation of chemotherapy in Cycle 2
Population: The population consisted of all participants who received chemotherapy, received a dose of study drug, had no protocol deviations and had complete data. Participants were grouped into 2 cohorts based on type of chemotherapy received.
Measure: Number; unit: Percentage of Participants
Groups:
- Fosaprepitant 150 mg: AC-like Chemotherapy: Women with breast cancer receiving AC-like chemotherapy receive fosaprepitant 150 mg administered IV on Day 1 of Cycle 2 of chemotherapy
- Fosaprepitant 150 mg: CT Chemotherapy: Women with gynecological cancer receiving CT chemotherapy receive fosaprepitant 150 mg administered IV on Day 1 of Cycle 2 of chemotherapy
Arm/Group | Fosaprepitant 150 mg: AC-like Chemotherapy | Fosaprepitant 150 mg: CT Chemotherapy
Number analyzed (Participants) | 61 | 40
Percentage of Participants | 62.30 | 50.00

3. Secondary Outcome: Percentage of Participants With a Complete Response During Cycle 2 of Chemotherapy
Description: A complete response is defined as no vomiting/no retching episodes and no use of rescue medication during the 120 hours following initiation of chemotherapy. The percentage of participants with a complete response during Cycle 2 of chemotherapy was calculated.
Time Frame: Up to 120 hours following initiation of chemotherapy in Cycle 2
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 101
Percentage of Participants | 21.78

4. Secondary Outcome: Functional Living Index - Emesis (FLIE) Total Score During Cycle 2 of Chemotherapy
Description: The FLIE Total Score is an 18-question quality-of-life questionnaire on the impact of nausea and vomiting (9 questions on nausea and 9 questions on vomiting) on daily life. Each question uses a visual analog scale (VAS) to rate the impact of nausea/vomiting from 1 to 7. FLIE Total Scores are calculated by summing the responses to the 18 questions and can range from 18-126 (18=a great deal of impairment, 126=no impairment), with a higher score indicating less impairment due to nausea and vomiting. "No Impact" on daily life was defined as a FLIE Total Score >108. Participants completed the FLIE questionnaire on the morning of Day 6 following initiation of chemotherapy in Cycle 2; their responses covered their experiences with nausea and vomiting over the previous 5 days.
Time Frame: From Day 1 (prior to initiation of chemotherapy in Cycle 2) to morning of Day 6 (up to ~120 hours following initiation of chemotherapy in Cycle 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 101
Score on a Scale
  Day 1 (prior to chemotherapy) | 92.90 (9.58)
  Day 6 | 80.50 (18.79)

5. Secondary Outcome: Percentage of Participants With No Significant Nausea During Cycle 2 of Chemotherapy
Description: Participants rated their degree of nausea in response to "How much nausea have you had over the last 24 hours?" using a 100-mm visual analog scale (VAS, 0=no nausea, 100=nausea as bad as it could be) on Days 2-6 following initiation of chemotherapy. No significant nausea was defined as VAS score <25 mm over the 24-120 hours following initiation of chemotherapy. The percentage of participants who experienced no significant nausea during Cycle 2 of chemotherapy was calculated.
Time Frame: From 24 to 120 hours following initiation of chemotherapy in Cycle 2
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 101
Percentage of Participants | 47.52

6. Secondary Outcome: Percentage of Participants Who Used No Rescue Medication During Cycle 2 of Chemotherapy
Description: Participants recorded any use of rescue medication for established nausea/vomiting in their daily diaries from initiation of chemotherapy infusion through the morning of Day 6. The percentage of participants who used no rescue medication during Cycle 2 of chemotherapy was calculated.
Time Frame: Up to 120 hours following initiation of chemotherapy in Cycle 2
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant 150 mg
Number analyzed (Participants) | 101
Percentage of Participants | 30.69

ADVERSE EVENTS:
Time Frame: Up to Day 18 after study drug administration (Up to 18 days)
Description: The Safety Population consists of all participants who received a dose of study drug. Participants with breast cancers and gynecological cancers were pooled for safety analysis.
Arm/Group | Fosaprepitant 150 mg
Serious Adverse Events (participants affected / at risk) | 6/111
Other Adverse Events (participants affected / at risk) | 64/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant 150 mg (N=111)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant 150 mg (N=111)
Constipation (Gastrointestinal disorders) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Eructation (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 18 (19)
Fatigue (General disorders) | 27 (27)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12)
Dizziness (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 18 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.